CLINICAL TRIAL: NCT02990663
Title: The Effect of Antihypertensive Medication Timing on Morbidity and Mortality: The "BedMed" RCT
Brief Title: The Effect of Antihypertensive Medication Timing on Morbidity and Mortality
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Innovates Health Solutions (Other); Alberta Health services (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BedMed Nov 30 2016
Record Dates: First submitted 2016-12-05; First posted 2016-12-13 (Estimated); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Hypertension
Keywords: Pragmatic; Primary Care; Chronotherapy; Administrative Data; Stroke; Myocardial Infarction; Congestive Heart Failure; Glaucoma; Dementia; Hip Fracture
MeSH Terms: conditions — Hypertension; Stroke; Myocardial Infarction; Heart Failure; Glaucoma; Dementia; Hip Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bedtime BP Meds (Experimental): Use of blood pressure lowering medication at bedtime
  Interventions: Other: Use of blood pressure lowering medication at bedtime
- Morning BP Meds (Active Comparator): Use of blood pressure lowering medication in the morning
  Interventions: Other: Use of blood pressure lowering medication in the morning

INTERVENTIONS:
Other: Use of blood pressure lowering medication at bedtime — Blood pressure lowering medications will be switched (one at a time as tolerated) to bedtime, or maintained at bedtime if already taken at that time. All decisions related to which, and how many, medications to switch are at the discretion of the care provider.
  Arms: Bedtime BP Meds
Other: Use of blood pressure lowering medication in the morning — Blood pressure lowering medications will be switched (one at a time as tolerated) to morning, or maintained in the morning if already taken at that time. All decisions related to which, and how many, medications to switch are at the discretion of the care provider.
  Arms: Morning BP Meds

SUMMARY:
High blood pressure is common and its presence increases the risk of cardiovascular mortality and morbidity (most notably stroke, myocardial infarction, and congestive heart failure). Given blood pressure is normally higher during the day than it is overnight, blood pressure lowering medications are traditionally taken in the morning. However a randomized trial of 2156 Spanish hypertension patients published in 2010 ("MAPEC"), suggests a large (61%) reduction in mortality and cardiovascular morbidity if such medications are instead taken at bedtime. This degree of benefit far exceeds other established methods of cardiovascular risk reduction - and such a surprisingly large effect requires independent confirmation for practice to change. BedMed is a pragmatic randomized controlled trial facilitated by over 400 Canadian family physician members of the Pragmatic Trials Collaborative. During the conduct of this trial consenting hypertensive primary care patients, already established on one or more antihypertensive medications, will be randomized to either morning or bedtime antihypertensive use. Patient oriented trial outcomes evaluating both potential benefits and harms will be drawn largely from administrative health data that is routinely collected on all residents of Canada's publicly funded health care system. This trial is being conducted in 5 Canadian provinces and will continue to collect data until late 2023, at which point more than 255 primary outcome events are anticipated.

DETAILED DESCRIPTION:
THE OPPORTUNITY BEDTIME PRESCRIBING MIGHT PROVIDE: Blood pressure normally exhibits a circadian rhythm with relatively lower pressures during sleep.(Ref 1) Lack of this sleep time "dip" correlates strongly with adverse cardiovascular events and BP correlates most strongly with such events when measured at night (i.e. during sleep).(Ref 2-5) Motivated by such observations, Spanish researchers studied the effect of taking BP medication at BEDTIME (when the effect on nighttime BP would be greatest) versus conventional morning use, when most BP medications are taken. The results of this study (the MAPEC trial) were striking.(Ref 6) Over a median 5.6 years follow-up, adverse cardiovascular events occurred in 187 of 1084 subjects taking BP medication in the morning but only 68 of 1072 subjects who took their BP medication at bedtime (relative risk 0.39, 95%CI [0.29-0.51], p < 0.001). This 61% reduction in adverse events was similar for all individual components of the primary outcome (including death from all causes, stroke, MI, new angina pectoris, CHF and retinal artery occlusions). If true, a switch to bedtime prescribing would have more impact on the health of hypertensive patients than whether high BP is treated at all. However extraordinary claims require extraordinary evidence - independent replication of such surprising findings is needed for widespread practice change to occur.

BEDMED: The BedMed trial is a pragmatic primary care trial intended to verify whether bedtime antihypertensive use, as compared to conventional morning use, reduces major adverse cardiovascular events. It is designed as an adaptive randomized registry trial within community primary care and draws both trial outcomes and baseline covariates from provincial administrative claims data (vital statistics, hospital separations, physician services, prescription dispenses, laboratory data). BedMed is government funded/facilitated, and has over 400 volunteer primary care providers recruiting participants in 5 Canadian provinces (Alberta, British Columbia, Saskatchewan, Manitoba, and Ontario). It was originally intended that the trial would continue until 406 primary outcome events were observed, however funding will expire before this occurs. As a result, BedMed will continue to recruit participants until early 2022 and complete data collection in late 2023, at which time more than 255 primary outcome events are anticipated (based on blinded observation of total events gathered at the end of 2021). The trial relies heavily on a collaboration between the volunteer family physicians of the Pragmatic Trials Collaborative (www.PragmaticTrials.ca) who will recruit for the trial and the Alberta SPOR Support Unit's Data Platform - which will facilitate accessing and analyzing the relevant administrative databases from multiple provinces (http://www.aihealthsolutions.ca/initiatives-partnerships/spor/).

DIURETIC SUB-STUDY: The "adaptive" element of the BedMed trial design refers to an interim examination of bedtime diuretic tolerance. Although it is commonly believed that diuretics can't be taken at bedtime without inducing unwanted nocturia, the sparse evidence in the literature suggests this may not be the case.(Ref 7,8) Rather than excluding patients whose only medication is a diuretic the investigators will instead initially include such patients and evaluate bedtime diuretic tolerance early on in the trial to determine whether or not such patients should continue to be enrolled. Specifically, upon allocating to bedtime dosing 203 patients whose only BP medication is an AM diuretic, the investigators will analyze 6-week compliance to bedtime allocation for all participants with a single morning BP medication (of all types). If diuretic compliance is worse, the "adaptive" trial design will exclude enrolment of additional patients whose only BP medication is a diuretic. The BedMed investigators will report on bedtime diuretic tolerance separate from (and in advance of) the main BedMed analysis.

INTERIM SAFETY ANALYSIS: An independent data safety monitoring board (DSMB) organized and chaired by Jim Wright (Cochrane Hypertension Review Group Coordinating Editor) is expected to review all data in March 2022, at which time approximately 150-160 primary outcome events are expected. If p is ≤ 0.001 for benefit (the Haybittle-Peto boundary - recommended to reduce the chance of stopping too early and magnifying benefit), or if p is ≤ 0.05 for harm, the DSMB will apply clinical judgement and make recommendations to the steering committee on whether the trial should stop early.

ELIGIBILITY:
Inclusion Criteria:

1. Hypertension diagnosis as assigned by a physician or nurse practitioner
2. ≥ 1 blood pressure medication taken once daily, or primary care provider willing to convert ≥ 1 blood pressure medication to once daily
3. Community dwelling (i.e. not residing in a nursing home; assisted living permitted)

Exclusion Criteria:

1. Palliative (as per primary care provider's judgement)
2. Unable to provide informed consent (as per primary care provider's judgement)
3. Personal history of glaucoma or use of glaucoma medications
4. Sleep disrupting shift work (more than 3 shifts/month during participant's regular sleeping hours)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3357 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events | Through study completion, an average of 4 years
  First occurrence of either death (all-cause), or hospitalization or emergency department visit for acute coronary syndrome / MI, congestive heart failure, or stroke.

SECONDARY OUTCOMES:
All-cause mortality | Through study completion, an average of 4 years
  Death from any cause.
Acute coronary syndrome | Through study completion, an average of 4 years
  Hospitalization or ER visit for acute coronary syndrome or MI.
CHF Hospitalization | Through study completion, an average of 4 years
  Hospitalization or ER visit for congestive heart failure.
Stoke | Through study completion, an average of 4 years
  Hospitalization or ER visit for stroke (excludes TIA).
All-cause hospitalization | Through study completion, an average of 4 years
  Hospitalization or ER visit for any cause
Long term care admission | Through study completion, an average of 4 years
  Newly admitted to a nursing home or assisted living facility as primary residence
New glaucoma diagnosis | Through study completion, an average of 4 years
  First-ever glaucoma diagnosis
Non-vertebral fracture | Through study completion, an average of 4 years
  Fracture of any bone other than the vertebra of the back or neck
Cognitive decline | 18 months
  Cognitive performance worsening by 2 or more points compared to baseline, as measured by the Short Blessed Test

OTHER OUTCOMES:
Acute care costs | Through study completion, an average of 4 years
  Acute care costs (derived from each admission's resource intensity weight and length of stay)
Total cost of care | Through study completion, an average of 4 years
  Acute care costs + medication costs + physician billings
Self-reported Overall Health Score | 1 year
  As measured by the EQ-5D-5L
Light-headedness | Through study completion, an average of 4 years
  Self-reported light-headedness or feeling "faint" without loss or consciousness in the prior month - yes / no. (Asked at 6-weeks, 6 months, and every 6 months)
Syncope | Through study completion, an average of 4 years
  Self-reported fainting (loss of consciousness) in the prior month - yes / no. (Asked at 6-weeks, 6 months, and every 6 months)
Falling | Through study completion, an average of 4 years
  Self-reported falling in the prior month - yes / no. (Asked at 6-weeks, 6 months, and every 6 months)
Nocturnal and daytime blood pressure | 6 months
  302 subjects will undergo 24-hour BP monitoring after 6 months to determine differences in blood pressure between groups.
Self-reported worsening of vision | Through study completion, an average of 4 years
  Vision self-reported as "much worse" compared to the last follow-up at any point, or "slightly worse" than the last follow-up, on 2 or more occasions (Note: vision is reported at 6-weeks, 6-months, and every 6-months, as either "unchanged", "slightly worse", or "much worse" than the last follow-up)
New impairment consistent with dementia | Through study completion, an average of 4 years
  Short Blessed Test score newly 10 or greater at 18-month assessment, or new physician administrative claims diagnosis of dementia at any point during follow-up
Hip fracture | Through study completion, an average of 4 years
  Any break of the hip joint or femoral neck
Nocturia frequency | 6-months
  Self-reported change from baseline in the number of overnight urinations per week (at 6-weeks and 6-months)
Nocturia burden | 6-months
  Self-reported nocturia burden in the prior month, recorded as no nocturia, or nocturia that is "no problem", "minor problem", or "major problem" (at 6-weeks and 6-months)
Adherence to medication timing allocation | 6-months
  Proportion of BP medication doses taken at the allocated time at 6-months (twice daily medications being considered as ½ dose in the AM and ½ dose in the PM for this calculation)

CONTACTS AND LOCATIONS:
Overall Officials: Scott R Garrison, MD, PhD, Principal Investigator — University of Alberta
Locations (5):
- Canada (5):
  - University of Alberta, Edmonton, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - University of Manitoba, Winnipeg, Manitoba
  - University of Toronto, Toronto, Ontario
  - University of Saskatchewan, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: Yes
Upon completion of all planned studies related to this project, anonymized patient level data for all outcomes and baseline characteristics will be made available in the form of a downloadable spreadsheet accessed through the Pragmatic Trials Collaborative's website (www.PragmaticTrials.ca)

REFERENCES:
- [Background] Veerman DP, Imholz BP, Wieling W, Wesseling KH, van Montfrans GA. Circadian profile of systemic hemodynamics. Hypertension. 1995 Jul;26(1):55-9. doi: 10.1161/01.hyp.26.1.55. PMID 7607733
- [Background] Clement DL, De Buyzere ML, De Bacquer DA, de Leeuw PW, Duprez DA, Fagard RH, Gheeraert PJ, Missault LH, Braun JJ, Six RO, Van Der Niepen P, O'Brien E; Office versus Ambulatory Pressure Study Investigators. Prognostic value of ambulatory blood-pressure recordings in patients with treated hypertension. N Engl J Med. 2003 Jun 12;348(24):2407-15. doi: 10.1056/NEJMoa022273. PMID 12802026
- [Background] Verdecchia P, Porcellati C, Schillaci G, Borgioni C, Ciucci A, Battistelli M, Guerrieri M, Gatteschi C, Zampi I, Santucci A, Santucci C, Reboldi G, et al. Ambulatory blood pressure. An independent predictor of prognosis in essential hypertension. Hypertension. 1994 Dec;24(6):793-801. doi: 10.1161/01.hyp.24.6.793. PMID 7995639
- [Background] Ben-Dov IZ, Kark JD, Ben-Ishay D, Mekler J, Ben-Arie L, Bursztyn M. Predictors of all-cause mortality in clinical ambulatory monitoring: unique aspects of blood pressure during sleep. Hypertension. 2007 Jun;49(6):1235-41. doi: 10.1161/HYPERTENSIONAHA.107.087262. Epub 2007 Mar 26. PMID 17389258
- [Background] Fagard RH, Celis H, Thijs L, Staessen JA, Clement DL, De Buyzere ML, De Bacquer DA. Daytime and nighttime blood pressure as predictors of death and cause-specific cardiovascular events in hypertension. Hypertension. 2008 Jan;51(1):55-61. doi: 10.1161/HYPERTENSIONAHA.107.100727. Epub 2007 Nov 26. PMID 18039980
- [Background] Hermida RC, Ayala DE, Mojon A, Fernandez JR. Influence of circadian time of hypertension treatment on cardiovascular risk: results of the MAPEC study. Chronobiol Int. 2010 Sep;27(8):1629-51. doi: 10.3109/07420528.2010.510230. PMID 20854139
- [Background] Rembratt A, Norgaard JP, Andersson KE. Nocturia and associated morbidity in a community-dwelling elderly population. BJU Int. 2003 Nov;92(7):726-30. doi: 10.1046/j.1464-410x.2003.04467.x. PMID 14616455
- [Background] Asplund R. Nocturia in relation to sleep, health, and medical treatment in the elderly. BJU Int. 2005 Sep;96 Suppl 1:15-21. doi: 10.1111/j.1464-410X.2005.05653.x. PMID 16083452
- [Derived] Garrison SR, Bakal JA, Kolber MR, Korownyk CS, Green LA, Kirkwood JEM, McAlister FA, Padwal RS, Lewanczuk R, Hill MD, Singer AG, Katz A, Kelmer MD, Gayayan A, Campbell FN, Vucenovic A, Archibald NR, Yeung JMS, Youngson ERE, McGrail K, O'Neill BG, Greiver M, Manca DP, Kraut RY, Wang T, Manns BJ, Mangin DA, MacLean C, McCormack J, Wong ST, Norris C, Allan GM. Antihypertensive Medication Timing and Cardiovascular Events and Death: The BedMed Randomized Clinical Trial. JAMA. 2025 Jun 17;333(23):2061-2072. doi: 10.1001/jama.2025.4390. PMID 40354045
- [Derived] Garrison SR, Kelmer M, Korownyk T, Kolber MR, Allan GM, Bakal J, Singer A, Katz A, Mcalister F, Padwal RS, Lewanczuk R, Hill MD, McGrail K, O'Neill B, Greiver M, Manca DP, Mangin D, Wong ST, Kirkwood JEM, McCormack JP, Yeung JMS, Green L. Tolerability of bedtime diuretics: a prospective cohort analysis. BMJ Open. 2023 Jun 6;13(6):e068188. doi: 10.1136/bmjopen-2022-068188. PMID 37280022
- [Derived] Garrison SR, Kolber MR, Allan GM, Bakal J, Green L, Singer A, Trueman DR, McAlister FA, Padwal RS, Hill MD, Manns B, McGrail K, O'Neill B, Greiver M, Froentjes LS, Manca DP, Mangin D, Wong ST, MacLean C, Kirkwood JE, McCracken R, McCormack JP, Norris C, Korownyk T. Bedtime versus morning use of antihypertensives for cardiovascular risk reduction (BedMed): protocol for a prospective, randomised, open-label, blinded end-point pragmatic trial. BMJ Open. 2022 Feb 24;12(2):e059711. doi: 10.1136/bmjopen-2021-059711. PMID 35210352
- See also: The Pragmatic Trials Collaborative — http://pragmatictrials.ca/